CLINICAL TRIAL: NCT05362682
Title: Effectiveness Evaluation of the Sinopharm Vaccine in the Dondo District in Mozambique
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: International Vaccine Institute (Other)
Collaborators: The Coalition for Epidemic Preparedness Innovations (CEPI) (Unknown); Instituto Nacional de Saúde, Mozambique (Other Government); University of Antananarivo (Unknown); International Centre for Diarrhoeal Disease Research, Bangladesh (Other); Harvard University (Other); Heidelberg University (Other)
Responsible Party: Sponsor
Other Study IDs: IVI-ECOVA-03
Record Dates: First submitted 2022-05-02; First posted 2022-05-05 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Sars-CoV-2 Infection
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case
  Interventions: Other: Sinopharm Vaccine
- Test Negative Control
  Interventions: Other: Sinopharm Vaccine

INTERVENTIONS:
Other: Sinopharm Vaccine — Sinopharm Vaccine will be administered by the Govt as part of COVID-19vaccination campaign

SUMMARY:
Three complementary activities will be implemented:1) Baseline and repeat census of the catchment population; described in a separate protocol (IVI-ECOVA-03-WS1); 2) Enhanced surveillance for COVID-19 disease, and 3) AEFI-enhanced surveillance. The mass vaccination campaign will be conducted by the Government and is not part of this protocol.

ELIGIBILITY:
Inclusion Criteria:

1. They resided in the study area at the time of mass immunization with the Sinopharm vaccine; and
2. They are at least 18 years of age during first round of mass vaccination.
3. Their onset of symptoms was <10 days prior to testing.
4. For each selected PCR test-positive case, we will select up to 3 test-negative controls from generally eligible subjects, matched to each case by age on the date of testing, sex, and calendar date of testing + 3 days.

Exclusion Criteria:

1. We will exclude subjects for selection as controls if they have had a positive test result within the following 21 days
2. Any Participant not matching the inclusion criteria mentioned above.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be conducted in the Dondo District. For surveillance the catchment area will include participants from Dondo Sede and Mafambisse administrative posts. The participant will come for screening in the following health facilities; Dondo, Baptista, Mandruzi, Canhandula, Samora Machel) and in Mafambisse (Mafambisse and Bloco Nove) and at the community level, the study will involve walk-throughs for COVID-19 testing.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2022-02-24 (Actual); Primary Completion 2024-02-28 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Protection conferred by two completed doses of Sinopharm vaccine against confirmed COVID-19 disease | 2 years
  Protection conferred by two completed doses of Sinopharm vaccine against RT-PCR-confirmed COVID-19 disease measured as the reduction in risk in adults who received two completed doses of the vaccine compared to those who are not vaccinated.

SECONDARY OUTCOMES:
Evaluate the effectiveness of two completed doses of the Sinopharm vaccine against severe SARS-CoV-2 infection | 2 years
  Evaluate the effectiveness of two completed doses of the Sinopharm vaccine against RT-PCR confirmed severe SARS-CoV-2 infection

CONTACTS AND LOCATIONS:
Locations (1):
- Dondo Health Facility, Dondo, Mozambique

IPD SHARING:
Plan to Share IPD: No